CLINICAL TRIAL: NCT00967785
Title: A Phase I Study of MozobilTM in the Treatment of Patients With WHIMS
Brief Title: A Phase I Study of Mozobil in the Treatment of Patients With WHIMS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090200; 09-I-0200
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2025-08-11

CONDITIONS: Leukopenia; Neutropenia; Infections; Warts; Myelokathexis
Keywords: Neutropenia; Hypogammaglobulinemia; Myelokathexis; Warts; Immunodeficiency
MeSH Terms: conditions — Leukopenia; Neutropenia; Infections; Warts; Agammaglobulinemia; Immunologic Deficiency Syndromes | interventions — plerixafor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Active Comparator): neutropenia and infections
  Interventions: Drug: Mozobil (TM)

INTERVENTIONS:
Drug: Mozobil (TM) — twice daily subcutaneous injection or via continuous subcutaneous infusion

SUMMARY:
Background:

* WHIMS (Warts, Hypogammaglobulinemia, Infections, and Myelokathexis Syndrome) is caused by various genetic changes that increase the activity of the chemokine receptor, CXCR4. Excessive function of this receptor causes mature neutrophils (part of the white blood cells) to be retained within the bone marrow rather than being released to the blood and is one of the causes of severe inherited neutropenia (low white blood counts). In neutropenia, the body is less able to fight off infection. Patients with WHIMS usually are at risk for skin, soft tissue, sinus, and lung infections, which can result in loss of hearing, teeth, and lung function.
* Current treatment for WHIMS consists of regular injections of a white blood cell growth stimulating medication called granulocyte colony stimulating factor (G-CSF), and supplemental immunoglobulin (antibody). These therapies are expensive, nonspecific, have significant side effects and toxicities, and do not fully correct all problems, especially warts and cancers related to human papillomavirus (HPV).
* A drug called Mozobil has been approved for use in combination with G-CSF to increase the number of stem cells that can be collected prior to bone marrow transplantation. Mozobil may offer a specific and well-tolerated new treatment for WHIMS and other syndromes characterized by neutropenia.

Objectives:

* To evaluate whether Mozobil is safe and effective to treat neutropenia (low white blood cell count) in patients with WHIMS.
* To determine an appropriate treatment dose of Mozobil, within currently approved dosage levels.

Eligibility:

- Individuals between 18 and 75 years of age who have been diagnosed with WHIMS and have a history of severe infections.

Design:

* Potential participants will undergo a screening with a medical history, physical examination, questionnaire, heart and lung function scans, and blood and urine samples. Tests will also be done for hepatitis B and C virus, and human immunodeficiency virus (HIV) that causes acquired immunodeficiency syndrome (AIDS), as well as to check neutrophil function.
* Patients who are being treated with G-CSF will stop injections for 2 days before being admitted to the National Institutes of Health (NIH) Clinical Center.
* Patients may participate in a Dose Escalation study and receive increasing doses of Mozobil over 5 days of treatment until their white blood cell count improves sufficiently or the maximum approved dose is reached. Blood samples will be taken regularly throughout the treatment process. Patients will then receive an additional dose of Mozobil at the maximum approved dose or the dose sufficient to cause improvement, before restarting the G-CSF injections.
* Patients may also participate in a long-term Chronic Dosing study and receive Mozobil once or twice a day for up to a maximum of 60 months.

DETAILED DESCRIPTION:
Mozobil (TM) (plerixafor injection, Genzyme/Sanofi) is a Food and Drug Administration approved medication to mobilize CD34+ hematopoietic stem cells prior to apheresis and use in autologous transplantation in non-Hodgkin lymphoma and multiple myeloma when used in conjunction with granulocyte-colony stimulating factor (G-CSF). The drug s mechanism of action is the specific and reversible inhibition of the chemokine receptor, CXCR4, expressed on CD34+ cells and other leukocytes. This inhibition interferes with the binding of stromal cell derived factor-1 (SDF-1), which is constitutively expressed on bone marrow stromal cells and appears to cause direct and indirect cellular adhesive interactions. Severe congenital neutropenia is a rare inherited disorder in which the affected individuals develop chronic or cyclical neutropenia with circulating counts below 500 cells/microliter blood. This disorder may result from a variety of genetic defects in progenitor- or neutrophil-expressed genes such as elastase, CXCR4, G6PC3, etc. Myelokathexis is the abnormal retention of mature leukocytes in the bone marrow and is seen in some types of severe chronic neutropenia such as warts, hypogammaglobulinemia, infections, and myelokathexis syndrome (WHIMS). WHIMS is a rare primary immunodeficiency, which is known to be caused by mutations that enhance CXCR4 signaling. Our hypothesis is that Mozobil(TM) can be used safely to partially block CXCR4 and treat neutropenia resulting from myelokathexis at doses considerably lower than that being used for CD34+ cell mobilization. This new treatment could also improve other aspects of the disease such as frequent infections, warts, and hypogammaglobulinemia. To test this hypothesis, we propose this trial of Mozobil (TM) in adults with WHIMS, examining safety and absolute neutrophil count as the primary endpoint. Mozobil is injected subcutaneously and will be injected via syringes (up to 84 months) or via an infusion pump (pilot trial of up to 10 subjects for a 24-month period).

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following inclusion criteria must be met for a subject to be enrolled in this study:

* Clinical diagnosis of WHIMS and documented severe infection
* Must be greater than or equal to 18 and less than or equal to 75 years of age
* Willingness to interrupt medications to raise the white count (WBC) such as G-CSF or GM-CSF for at least 2 days before and while on the study drug
* Must not be pregnant or breastfeeding
* Must have a personal physician
* Must be willing to provide blood, plasma, serum, and DNA samples for storage
* Subjects must agree not to become pregnant or to impregnate a female. If of childbearing potential, must agree to consistently use two types of contraception throughout study participation. Acceptable forms of contraception include the following:

  1. Condoms, male or female, with or without a spermicide
  2. Diaphragm or cervical cap with spermicide
  3. Intrauterine device
  4. Contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
  5. Male partner has previously undergone a vasectomy for which there is documentation of aspermatogenic sterility

EXCLUSION CRITERIA:

If any of the following exclusion criteria are met, a subject will not be enrolled in this study:

* Absence of a diagnosis of WHIMS
* Patient is less than 18 years old
* Absence of a documented history of severe infection
* Neutropenia due to maturation defects in the myeloid lineage or that the PI feels is unlikely to benefit from this medication
* Pregnant women or breastfeeding
* History of serious cardiac arrhythmia or cardiac defects that make such more likely
* Renal failure (calculated creatinine clearance [CrCl] <15 mL/min or requiring dialysis)
* Signs or symptoms of active microbial infection at the time of study entry.
* Any condition that, in the investigator s opinion, places the patient at undue risk by participating in the study
* Unwillingness to undergo testing or procedures associated with this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | Duration of treatment, up to 7 years
  No incident of grade 3/4 toxicities.
Increase ANC | Duration of treatment, up to 7 years.
  Average ANC > 250 and > twice baseline level.

SECONDARY OUTCOMES:
reduced HPV lesions | duration of treatnebt, up to 6 years.
  photographs demonstrating reduced warts, after extended period of treatment.
Increase Leucocytes | prior to and after study drug
  statistically significant increase leucocyte after drug injection.

CONTACTS AND LOCATIONS:
Overall Officials: David H McDermott, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDermott DH, Majumdar S, Velez D, Cho E, Li Z, Gao JL, Grieco MC, Lawrence MG, Silva SL, Castelo-Soccio LA, Follmann D, Murphy PM. Continuous Infusion of the CXCR4 Antagonist Plerixafor for WHIM Syndrome. medRxiv [Preprint]. 2025 Apr 22:2025.04.19.25325865. doi: 10.1101/2025.04.19.25325865. PMID 40330596
- [Derived] Broxmeyer HE. A WHIM satisfactorily addressed. Blood. 2014 Apr 10;123(15):2286-8. doi: 10.1182/blood-2014-02-557579. PMID 24723677
- [Derived] McDermott DH, Liu Q, Velez D, Lopez L, Anaya-O'Brien S, Ulrick J, Kwatemaa N, Starling J, Fleisher TA, Priel DA, Merideth MA, Giuntoli RL, Evbuomwan MO, Littel P, Marquesen MM, Hilligoss D, DeCastro R, Grimes GJ, Hwang ST, Pittaluga S, Calvo KR, Stratton P, Cowen EW, Kuhns DB, Malech HL, Murphy PM. A phase 1 clinical trial of long-term, low-dose treatment of WHIM syndrome with the CXCR4 antagonist plerixafor. Blood. 2014 Apr 10;123(15):2308-16. doi: 10.1182/blood-2013-09-527226. Epub 2014 Feb 12. PMID 24523241
- [Derived] McDermott DH, Liu Q, Ulrick J, Kwatemaa N, Anaya-O'Brien S, Penzak SR, Filho JO, Priel DA, Kelly C, Garofalo M, Littel P, Marquesen MM, Hilligoss D, Decastro R, Fleisher TA, Kuhns DB, Malech HL, Murphy PM. The CXCR4 antagonist plerixafor corrects panleukopenia in patients with WHIM syndrome. Blood. 2011 Nov 3;118(18):4957-62. doi: 10.1182/blood-2011-07-368084. Epub 2011 Sep 2. PMID 21890643
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-I-0200.html